CLINICAL TRIAL: NCT02760771
Title: Transfemoral Transcatheter Aortic Valve Implantation With or Without Predilation of the Aortic Valve (EASE-IT TF)
Acronym: EASE-IT-TF
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: EASE-IT-TF
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Aortic Stenosis
Keywords: THV (trans-catheter heart valve); severe aortic stenosis; pre-dilation; rapid pacing; BAV (balloon artery valvuloplasty
MeSH Terms: conditions — Aortic Valve Stenosis; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with BAV: patients undergoing transfemoral trans-catheter aortic valve implantations (TF-TAVI) with predilation of the aortic valve
  Interventions: Other: with BAV
- without BAV: patients undergoing transfemoral trans-catheter aortic valve implantations (TF-TAVI) without predilation of the aortic valve
  Interventions: Other: without BAV

INTERVENTIONS:
Other: with BAV — balloon dilation of the aortic valve prior to implantation of the THV
  Groups: with BAV
Other: without BAV — no balloon dilation of the aortic valve prior to implantation of the THV
  Groups: without BAV

SUMMARY:
Prior to the deployment of transcatheter heart valves (THV), balloon aortic valvuloplasty (BAV) is often performed under rapid right ventricular pacing (burst >180 bpm) with the induction of a functional cardiac arrest for up to 30 seconds. Aortic valve predilation aims at facilitating the crossing of the aortic annulus, accurate valve positioning and does also provide information on the anatomy of the valve complex. However, BAV has been shown to have a number of potentially detrimental effects.

There is limited experience for the balloon expandable Edwards THV on the need for predilation (BAV). Experience so far has only been documented from smaller, uncontrolled case series.

The investigators aim to document the incidence of several kinds of complications in a large, multicenter registry / prospective controlled cohort study to identify associations between patient related variables and outcomes.

DETAILED DESCRIPTION:
Aortic valve predilation aims at facilitating the crossing of the aortic annulus, accurate valve positioning and does also provide information on the anatomy of the valve complex. However, BAV has been shown to have a number of potentially detrimental effects, such as:

* Functional cardiac arrest induced by rapid pacing leads to transient coronary, cerebral, and renal ischemia.
* In patients with a reduced left ventricular ejection fraction (LVEF), prolonged cardiac depression after rapid pacing is observed and may result in hemodynamic failure and systemic inflammatory response syndrome (SIRS). Both are associated with a high periprocedural mortality.
* BAV has been identified as a major source of thrombotic and valvular material, thus increasing the risk for coronary obstruction with subsequent myocardial infarction and/or stroke.
* The local trauma in the left-ventricular outflow tract caused by BAV may potentially contribute to aortic root rupture.

The investigators aim to document the incidence of cerebrovascular complications, paravalvular leakage and operative outcomes in a large, multicenter registry / prospective controlled cohort study to identify associations between patient related variables and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Males or females
* At least 18 years of age

Exclusion Criteria:

* Logistic EuroSCORE I >40%
* Mitral or tricuspid valvular insufficiency (> grade II)
* Previous aortic valve replacement
* Uncontrolled atrial fibrillation
* Left ventricular or atrial thrombus by echocardiography
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Patients with mobile structures on the leaflets
* Need for a cerebral protection device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for transfemoral transcatheter valve implantation with commercially available Edwards Transcatheter Heart Valves.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Combination of all-cause mortality, stroke, non-fatal myocardial infarction, acute kidney injury, or pacemaker implantation | within 30 days after TAVI

SECONDARY OUTCOMES:
All-cause mortality | within 30 days after TAVI
Stroke | within 30 days after TAVI
Non-fatal myocardial infarction | within 30 days after TAVI
pacemaker implantation | within 30 days after TAVI
acute kidney injury | within 30 days after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schymick, MD, Principal Investigator — Städtisches Klinikum Karlsruhe; David Wendt, PD MD, Principal Investigator — Westdeutsches Herzzentrum Essen
Locations (1):
- Medizinische Klinik IV, Städtisches Klinikum Karlsruhe, Karlsruhe, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schymik G, Rudolph T, Jacobshagen C, Rothe J, Treede H, Kerber S, Frank D, Sykorova L, Okamoto M, Thoenes M, Deutsch C, Bramlage P, Butter C. Balloon-expandable transfemoral transcatheter aortic valve implantation with or without predilation: findings from the prospective EASE-IT TF multicentre registry. Open Heart. 2019 Oct 3;6(2):e001082. doi: 10.1136/openhrt-2019-001082. eCollection 2019. PMID 31673387
- [Derived] Butter C, Bramlage P, Rudolph T, Jacobshagen C, Rothe J, Treede H, Kerber S, Frank D, Seilerova L, Schymik G. Balloon expandable transcatheter aortic valve implantation via the transfemoral route with or without pre-dilation of the aortic valve - rationale and design of a multicentre registry (EASE-IT TF). BMC Cardiovasc Disord. 2016 Nov 15;16(1):223. doi: 10.1186/s12872-016-0390-4. PMID 27846807
- See also: registry on-line eCRF website — https://ippmed-easeittf.s4trials-europe.net